CLINICAL TRIAL: NCT03717207
Title: SGLT2-inhibitors Reduce the Cardiac Autonomic Neuropathy Dysfunction and Vaso-vagal Syncope Recurrence in Patients With Type 2 Diabetes Mellitus: the SCAN Study
Brief Title: Cardiac Autonomic Dysfunction in Diabetics Patients With Syncope
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, medical doctor, University of Campania Luigi Vanvitelli
Other Study IDs: 2210012018
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Syncope, Vasovagal
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type 2 diabetes mellitus (T2DM) patients under SGLT2-I therapy (SGLT2-I users): T2DM patients affected by vaso vagal syncope, and under SGLT2-I therapy. All these patients were in stable sinus rate before performing the HUT They performed a 24 hours ECG Holter to assess sinus rhythm, HR, HRV, and the MIBG myocardial scintigraphy before receiving a HUT.
  .
  Interventions: Other: ecg Holter,; Diagnostic Test: cardiac scintigraphy
- type 2 diabetes mellitus (T2DM) patients without SGLT2-I therapy (Non-SGLT2-I users): T2DM patients affected by vaso vagal syncope, and without SGLT2-I therapy. All these patients were in stable sinus rate before performing the HUT They performed a 24 hours ECG Holter to assess sinus rhythm, HR, HRV, and the MIBG myocardial scintigraphy before receiving a HUT.
  Interventions: Other: ecg Holter,; Diagnostic Test: cardiac scintigraphy

INTERVENTIONS:
Other: ecg Holter, — all patients before to perform an head up tilt test for syncope evaluation will be steadied by ecg Holter to assess heart rate, heart rate variability.
Diagnostic Test: cardiac scintigraphy — all patients before to perform an head up tilt test for syncope evaluation will receive a the 123I-MIBG, which is a norepinephrine analogous, to calculate the late heart-to-mediastinum ratio (H/Mlate) and washout rate (WR). Thus, we evaluated the H/Mlate as the index of global neuronal function due to norepinephrine uptake and the WR as the index of sympathetic tone.

SUMMARY:
Study hypothesis: cardiac autonomic dysfunction may affect vaso vagal syncope recurrences in type 2 patients with diabetes vs. patients without diabetes.

Background: vaso vagal syncope and its recurrences may be due to alterations in autonomic system function, that may be more frequent in diabetics. Heart rate variability (HRV) is a valid test to study sympathetic and vaso vagal tone dysfunction. However, in this study authors investigated the correlation between HRV alterations and diabetes in a population of patients affected by syncope, and classified as vaso vagal syncope by Head Up Tilt Test (HUT) exam. Secondly, authors assessed these alterations as causes of vaso vagal syncope recurring at 12 months of follow up in type 2 patients with diabetes under sodium-glucose transporter 2 inhibitors (SGLT2-inhibitors) vs. other hypoglycemic drugs .. Materials and Methods: In a multicenter study authors studied T2DM patients under SGLT2-I therapy (n 426) vs. those that did not receive the SGLT2-I therapy (n 2195), and affectede by vaso vagal syncope. All enrolled patients were in stable sinus rate before to perform ECG Holter, and the Head Up Tilt Test (HUT). However, before to perform the HUT all patients performed a 24 hours ECG Holter, to asses sinus rhythm , heart rate, and HRV. Then, these patients performed a 123I-metaiodobenzylguanidine (123I-MIBG) myocardial scintigraphy to assess cardiac autonomic dysfunction.

Moreover, authors performed a propensity score matching (PSM) analysis to evaluate 160 SGLT2-I users vs. 160 Non-SGLT2-I users' patients.

DETAILED DESCRIPTION:
Vaso vagal syncope recurrence is a relevant clinical problem (1). In fact, despite the vaso vagal syncope event is a transient loss of consciousness with rapid onset, short duration, and spontaneous complete recovery after the event, it may be complicated by physical injury (2). Conversely, the syncope recurrence rate is about 35%, and it causes a physical injury until the 29% (3). In addition, the vaso vagal syncope has a frequency between 15% and 39%, with annual number of episodes about 18.1-39.7 per 1000 patients, and an incidence of 6.2 per 1000 person-years, that grows up after 70 years of age with rate annual 19.5 per thousand individuals after 80 years (3). The patients with type 2 diabetes mellitus (T2DM) represent a percentage about the 30% of all the subjects with syncope (4). About the pathophysiology of syncope a central role is played by autonomic nervous system (5). To date, the autonomic nervous system regulates the hemodynamic stability by maintaining a stable blood pressure and heart rate under normal and abnormal physiologic conditions (5). Consequently, the dysfunction of this complex regulatory system, and of its interaction with sensor systems as baroreceptors, mechanoreceptors, chemoreceptors, may alter the vascular reactivity, leading to the clinical event and to future recurrences (5). Multiple factors affecting the autonomic system balance may trigger and cause a syncope event, as the result of an inappropriate response of the autonomic nervous system, with excessive vagal tone, and sympathetic tone withdrawal (2). In this setting, authors may note the diabetes as a common cause of autonomic system dysfunction (6). Moreover, T2DM may cause a severe form of autonomic system dysfunction affecting the cardiac autonomic regulation, and named as cardiac autonomic neuropathy (CAN), (6). Intriguingly, patients with diabetes experience a parasympathetic denervation, with an early augmentation of sympathetic tone, then leading to impaired heart rate variability, resting tachycardia, exercise intolerance, abnormal blood pressure regulation, and orthostatic hypotension (7). In addition, in T2DM there is a compensatory increase in the cardiac sympathetic tone in response to subclinical peripheral denervation (7). However, the T2DM may be seen as a relevant risk factor and a trigger to alter the autonomic system balance, and to cause vaso vagal syncope. In this context, the SGLT2-I are hypoglycemic drugs that might modulate the systemic and cardiac sympathetic dysfunction. On the other hand, the effects of the SGLT2-I therapy on the diabetic autonomic dysfunction and the vaso vagal syncope recurrence at follow up is not well established. Moreover, the recent studies cannot come to definitive conclusion about the impact of SGLT2-I on the vaso vagal syncope events, and about its future recurrences in patients with type 2 diebetes mellitus (T2DM). Conversely, heart rate variability (HRV) is a simple, reproducible and well-recognized method for evaluating sympatho vagal activity (8, 9). In this setting, the 123I-MIBG is an imaging exam to evaluate the cardiac autonomic dysfunction. Indeed, the 123I is an analogous of norepinephrine, and the entity of its myocardial captation is an index of cardiac innervation.

However, in this study authors evaluated the autonomic dysfunction as alteration in HRV, and 123I-MIBG, and its relevance to cause vaso vagal syncope, and the vaso vagal syncope recurrence in SGLT2-I users vs. Non-SGLT2-I users' patients with T2DM at 12 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of vaso vagal syncope, and left ventricle ejection fraction >55%.

Exclusion Criteria:

* patients with neuropathy, arterial hypertension, indications of heart failure and coronary heart disease or depression of left ventricle ejection fraction (LVEF < 55%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients with clinical history of vaso vagal syncope, as diagnosed by head up tilt test. These patients, aged between 18 and 75 years, received an ecg Holter before to perform head up tilt test evaluation. These patients presented with vaso vagal syncope in absence of neuropathy, arterial hypertension, heart failure and coronary heart disease or depression of left ventricle ejection fraction (LVEF < 55%).
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
syncope recurrence | 12 months.
  authors will report all syncope recurrences at 12 months of follow up in T2DM patients SGLT-I users vs. T2DM patients Non-SGLT2-I users.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, Massimo Massetti M, Rambaldi P, Gatta G, Cappabianca S, Sasso FC, Santamaria M, Volpicelli M, Ducceschi V, Signoriello G, Paolisso G, Marfella R. SGLT2-inhibitors reduce the cardiac autonomic neuropathy dysfunction and vaso-vagal syncope recurrence in patients with type 2 diabetes mellitus: the SCAN study. Metabolism. 2022 Dec;137:155243. doi: 10.1016/j.metabol.2022.155243. Epub 2022 Jun 19. PMID 35732222